CLINICAL TRIAL: NCT04703101
Title: Organ Preservation for Patients With Locally Advanced Rectal Adenocarcinoma: Evaluating the Efficacy of Short Course Radiation Therapy Followed by FOLFOX or CapeOX
Brief Title: Short Course Radiation Therapy and Combination Chemotherapy for the Treatment of Stage II-III Rectal Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: The Joseph Drown Foundation (Unknown); Natera, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-001156; NCI-2020-06479 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20-001156 (Other: UCLA / Jonsson Comprehensive Cancer Center)
Record Dates: First submitted 2021-01-07; First posted 2021-01-11 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-02

CONDITIONS: Locally Advanced Rectal Carcinoma; Rectal Adenocarcinoma; Stage II Rectal Cancer AJCC v8; Stage IIA Rectal Cancer AJCC v8; Stage IIB Rectal Cancer AJCC v8; Stage IIC Rectal Cancer AJCC v8; Stage III Rectal Cancer AJCC v8; Stage IIIA Rectal Cancer AJCC v8; Stage IIIB Rectal Cancer AJCC v8; Stage IIIC Rectal Cancer AJCC v8
MeSH Terms: conditions — Rectal Neoplasms | interventions — Capecitabine; Fluorouracil; dehydroftorafur; Radiotherapy, Intensity-Modulated; Leucovorin; Oxaliplatin

STUDY DESIGN:
Masking Description: Analysts blinded to patient outcome and sample order
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (IMRT, mFOLFOX6, CapeOX, TME) (Experimental): Patients undergo SCRT in the form of IMRT over 5 fractions daily for 5 consecutive days. Beginning 11-18 days after the last day of radiation therapy, patients receive either oxaliplatin IV and leucovorin IV on day 1 and fluorouracil IV on days 1-3 (mFOLFOX6) or oxaliplatin IV on day 1 and capecitabine PO BID on days 1-14 (CapeOX). Treatment with mFOLFOX6 repeats every 2 weeks for up to 8 cycles, and treatment with CapeOX repeats every 3 weeks for up to 6 cycles in the absence of disease progression or unacceptable toxicity. At 8-12 weeks after completion of all therapy, patients with residual tumor undergo TME. Patients with cCR undergo NOM.
  Interventions: Drug: Capecitabine; Drug: Fluorouracil; Radiation: Intensity-Modulated Radiation Therapy; Drug: Leucovorin; Drug: Oxaliplatin; Other: Quality-of-Life Assessment; Behavioral: Surveillance; Procedure: Total Mesorectal Excision

INTERVENTIONS:
Drug: Capecitabine — Given IV
  Other Names: Ro 09-1978/000; Xeloda
Drug: Fluorouracil — Given IV
  Other Names: 5 Fluorouracil; 5 Fluorouracilum; 5 FU; 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-Fu; 5FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
Radiation: Intensity-Modulated Radiation Therapy — Undergo IMRT
  Other Names: IMRT; Intensity Modulated RT; Intensity-Modulated Radiotherapy; Radiation, Intensity-Modulated Radiotherapy
Drug: Leucovorin — Given IV
  Other Names: Folinic acid
Drug: Oxaliplatin — Given IV
  Other Names: 1-OHP; Ai Heng; Aiheng; Dacotin; Dacplat; Diaminocyclohexane Oxalatoplatinum; Eloxatin; Eloxatine; JM-83; Oxalatoplatin; Oxalatoplatinum; RP 54780; RP-54780; SR-96669
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Behavioral: Surveillance — Undergo NOM
  Other Names: Epidemiology / Surveillance
Procedure: Total Mesorectal Excision — Undergo TME
  Other Names: TME

SUMMARY:
This phase I trial investigates how well short-course radiation therapy followed by combination chemotherapy works in treating patients with stage II-III rectal cancer. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Chemotherapy drugs, such as leucovorin, fluorouracil, oxaliplatin, and capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving short-course radiation therapy and combination chemotherapy may reduce the need for surgery and therefore improve quality of life.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Complete clinical response (cCR) rate of patients with clinical T3 and/or node-positive M0 rectal cancer being treated with short-course radiation therapy (SCRT) followed by 16 weeks of modified leucovorin, fluorouracil, and oxaliplatin (mFOLFOX)/capecitabine and oxaliplatin (CapeOX).

SECONDARY OBJECTIVES:

I. 1-year local recurrence free survival and 1-year progression free survival of the entire cohort, the cohort that initially undergoes non-operative management (NOM), and the cohort that initially undergoes total mesorectal excision (TME).

II. Physician-reported acute and late >= grade 3 toxicity rates. III. 1-year post-treatment patient health-related quality of life and anorectal function as per Patient Reported Outcomes Measurement and Information System (PROMIS).

IV. Explore how Signatera's residual disease test correlates with patient's cCR rates, local recurrence, progression-free, and overall survival rates.

V. Explore radiomics features from longitudinal diffusion weighted magnetic resonance imaging (MRI) (diffusion weighted imaging [DWI]) data and build a predictive model for treatment effect (complete response) in rectal cancer patients undergoing SCRT.

OUTLINE:

Patients undergo SCRT in the form of intensity-modulated radiation therapy (IMRT) over 5 fractions daily for 5 consecutive days. Beginning 11-18 days after the last day of radiation therapy, patients receive either oxaliplatin intravenously (IV) and leucovorin IV on day 1 and fluorouracil IV on days 1-3 (mFOLFOX6) or oxaliplatin IV on day 1 and capecitabine orally (PO) twice daily (BID) on days 1-14 (CapeOX). Treatment with mFOLFOX6 repeats every 2 weeks for up to 8 cycles, and treatment with CapeOX repeats every 3 weeks for up to 6 cycles in the absence of disease progression or unacceptable toxicity. At 8-12 weeks after completion of all therapy, patients with residual tumor undergo TME. Patients with cCR undergo NOM.

After completion of study treatment, patients who underwent NOM are followed up every 3 months for 2 years, then every 6 months for 3 years. TME patients are followed up every 3-6 months for 2 years, then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed rectal adenocarcinoma
* Patients must have stage II (cT3, cN0) or stage III (cT1-3, cN1-3) tumor as staged by MRI
* No evidence of metastatic disease
* Resectable primary lesion
* Karnofsky performance status (KPS) >= 70 or Eastern Cooperative Oncology Group (ECOG) 0-2
* Absolute neutrophil count (ANC) > 1.5 cell/mm^3
* Hemoglobin (Hgb) > 8.0 gm/dL
* Platelets (PLT) > 150,000/mm^3
* Total bilirubin < or equal to 1.5 x upper limit of normal
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < or equal to three times upper limit of normal
* If a woman is of childbearing potential, a negative serum pregnancy test must be documented prior to initiation of radiation therapy

Exclusion Criteria:

* Active treatment of a separate malignancy
* Distant metastatic disease as assessed by staging positron emission tomography (PET)/computed tomography (CT) or CT of the chest and abdomen within 6 weeks of starting radiation therapy
* Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields
* Pregnant and/or breastfeeding
* Medical/psychological contraindication to MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-02-11 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-10-15 (Estimated)

PRIMARY OUTCOMES:
Complete clinical response rate | Up to 5 years
  Kaplan-Meier analysis will be carried out and used to estimate for the entire cohort as well the non-operational management (NOM) and total mesorectal excision (TME) cohorts separately.

SECONDARY OUTCOMES:
Local recurrence-free survival | At 1 year
  Kaplan-Meier analysis will be carried out and used to estimate for the entire cohort as well the NOM and TME cohorts separately.
Progression-free survival | At 1 year
  Kaplan-Meier analysis will be carried out and used to estimate for the entire cohort as well the NOM and TME cohorts separately.
Incidence of adverse events | Up to 5 years
  Physician-reported acute and late >= grade 3 toxicity rates for the entire cohort will be graded according to Common Terminology Criteria for Adverse Events version 5.0.
Health-related quality of life | At 1 year
  Will be assessed by Patient Reported Outcomes Measurement and Information System and calculated and presented as a composite score. These scores will be calculated for the entire cohort as well as the NOM and TME cohorts separately.
Anorectal function | At 1 year
  Will be assessed by Patient Reported Outcomes Measurement and Information System and calculated and presented as a composite score. These scores will be calculated for the entire cohort as well as the NOM and TME cohorts separately.
Signatera's residual disease test | Up to 5 years
  Cox proportional hazards regression analysis will be used to assess the association of circulating tumor deoxyribonucleic acid with clinical response rates, local recurrent, progression-free, and overall survival rates.
Prediction of complete clinical response rate status by radiomics | Up to 5 years
  The relationship between complete clinical response as a binary variable and longitudinal radiomics features from a sequence of four diffusion weighted imaging data points will be assessed via a logistic regression model with a random effect term to account for within-subject correlation.

CONTACTS AND LOCATIONS:
Overall Officials: Ann Raldow, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States